CLINICAL TRIAL: NCT04614831
Title: Psoriasis and Beyond: A Worldwide Survey on the Understanding of Psoriatic Disease Among Patients With Psoriasis and Psoriatic Arthritis
Brief Title: A Worldwide Survey on the Understanding of Psoriatic Disease Among Patients With Psoriasis and Psoriatic Arthritis
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457A2023
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Plaque Psoriasis, Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Psoriasis and Psoriatic Arthritis: The study population consists of adults who self-report to have been diagnosed with psoriasis with or without concomitant psoriatic arthritis

SUMMARY:
The study is a Worldwide Survey on the Understanding of Psoriatic Disease among Patients with Psoriasis and Psoriatic Arthritis.

DETAILED DESCRIPTION:
This is a cross-sectional, quantitative online survey of patients with psoriasis with or without concomitant psoriatic arthritis. Following assessment of participant eligibility via a 5-minute online screener, the 25-minute internet-based survey will be conducted without any follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who self-report to have been diagnosed with Psoriasis or Psoriasis and Psoriatic Arthritis before or at the time of data collection
2. Patients 18 years of age or older at the time of data collection
3. Patients who did not participate in surveys regarding Psoriasis or Psoriatic Arthritis in the last 4 weeks
4. Body Surface Area (BSA) of >5 to <10, with psoriasis affecting sensitive and/or prominent body parts: face, palms, hands, fingers, genitals, soles of feet or nails or a BSA of 10 and above, when psoriasis was at its worst

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adults with self-reported Psoriasis and/or Psoriatic Arthritis. Screening questions will be used to determine the eligibility for each respondent to the survey.
Sampling Method: Non-Probability Sample
Enrollment: 4978 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
A web-based survey will be answered by the participants. Data collected for the analysis of the primary objective include validated patient-reported outcomes (such as DLQI), as well as responses to non-validated questions. | 1 Day of survey
  To assess patients' understanding of psoriasis and psoriatic arthritis as part of a systemic disease and the humanistic and physical burden of living with the condition.

SECONDARY OUTCOMES:
A web-based survey will be answered by the participants. The data collected for the analysis of the secondary objectives include validated tools (such as PAM-13), as well as responses to non-validated questions. | 1 Day of Survey
  To assess the patient's perceptions and attitudes related to the relationship with their physician, the patient journey through the healthcare system, as well as barriers to self-management, diagnosis, patient perceptions on biologics, treatment expectations, and satisfaction with care.

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Investigational Site, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No